CLINICAL TRIAL: NCT01364831
Title: Connection Between Sleep Quality and Duration and Performance in Young Athletes
Brief Title: Connection Between Sleep and Athletic Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wingate Institute (Other)
Responsible Party: Principal Investigator, Dr. Eyal Shargal, Professional director , The Ribstein Center for Sports Medicine and Research, Wingate Institute
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: WingateHC1
Record Dates: First submitted 2011-03-29; First posted 2011-06-02 (Estimated); Last update posted 2014-01-01 (Estimated); Status verified 2013-12

CONDITIONS: Quality Sleep Time; Athletic Performance
Keywords: sleep time; athletic performance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Sleep extension — Athletic performance evaluated at baseline and following about 1.5 hours of sleep extension

SUMMARY:
In the last few decades much knowledge has been accumulated on the connection between healthy, sufficient sleep and overall health, cognitive function, memory and job or school performance, motor vehicle accidents and work accidents. There has been growing awareness recently of the connection between physical activity and competitive sports performance, and the amount and quality of sleep. Despite the dearth of scientific studies, there is a constant effort to improve understanding in this field.

An appropriate procedure designed to evaluate the influence of the quality and amount of sleep on ability and athletic performance must fulfill a number of basic requirements:

1. Isolating the influence of components related to sleep homeostasis and factors relating to circadian rhythm.
2. Neutralizing as much as possible the influence of motivation on the evaluation - one must presumably include a significant competitive event (it is not always possible to do a simple extrapolation between physiological measurements and competitive performance).
3. Isolating and canceling as much as possible additional factors affecting performance, such as: home advantage, weather, injury and field conditions.

Athletic activity includes not just competitions but also training towards competitions, since it is difficult to control for influences of competitions and other occasional events, in this study the investigators focus on evaluation of the connection between sleep and athletic performance in training.

Towards the end of adolescence, youth are busy in multiple activities related to studies, social obligations and athletic activity. This is also the age they learn to drive. This is an age in which physiologically a person needs more sleep relative to at other ages (9.25 hours of sleep a day), and paradoxically due to the multiple obligations the amount of sleep is lower than needed.

Beyond the effect on mood, cognitive performance and memory, sleep deprivation causes far-reaching changes in multiple systems, such as:

Cardiovascular System:

* Many studies show that shortened sleep duration constitutes an independent cause of increased cardiac events.
* Resting heart rate and maximum heart rate decrease after 30 hours of sleep deprivation.

Respiratory System:

* Significant decline in respiratory function as measured by: FVC, Maximal voluntary ventilation, Maximal static inspiratory/expiratory pressures, Time to exhaustion with exercise, Peak O2 consumption, Peak CO2 production.
* Worsening of respiratory sleep disturbances.

Digestive System:

• Changes in food consumption accompanied by changes in body weight.

Neurophysiological System

• Disturbance of thermoregulation.

Endocrine System:

* Hormonal changes associated with hypothalamic-hypophyseal axis
* Influence on secretion of Ghrelin and leptin
* Influence on secretion of growth hormone.

In light of this, there is sound basis for the presumption that athletic performance is connected to these influences directly and indirectly.

The purpose of this study is to evaluate the connection between sleep quality and duration and athletic performance among young athletes living and training at the Sport-Gifted Centre at the Wingate Institute.

DETAILED DESCRIPTION:
Aim The purpose of this study is to evaluate the connection between sleep quality and duration and athletic performance among young athletes living and training at the Sport-Gifted Centre at the Wingate Institute.

Methods 50 athletes of the Sport-Gifted Centre at the Wingate Institute, ages 13-20, male and female, from the branches of triathlon and swimming. Participants and their parents will be asked to give informed consent.

The proposed study will have two stages:

1. Baseline assessment: In the first stage there will be an evaluation of sleep quality and duration of the athletes over the course of two weeks, in parallel their athletic performance will be evaluated using accepted measures such as: swimming times over set distances, running times over set distances, etc.
2. Assessment of intervention's effect of prolonging the duration of nighttime sleep on the athletic performance of the participants, using the same measures as above. This stage will take four weeks.

Stage 1:

Before beginning the study each participant will fill out a general health questionnaire.

Each participant will receive a Suunto heart monitor belt to sleep with for two weeks. Each participant will be asked to wear the belt before going to bed and take it off upon waking up in the morning. Heart rate data stored on the belts will be transferred each morning to a computer. Analysis of sleep architecture and duration over the course of the two weeks will be carried out using the HC1000P system from HypoCore Inc. (see attached documents). In addition average heart rate and maximal heart rate can be assessed while training at baseline by recording heart rate using the Suunto belts. Sleep data will be analyzed and each participant will receive a personalized analysis of his/her sleep. At this stage the investigators will evaluate the baseline characteristics of the participants including sleep duration, sleep efficiency, presence and duration of the different sleep stages, in particular slow wave sleep during which it is known a growth factor is released which is important for muscle recovery, times and durations of training sessions and athletic performance.

Evaluation of athletic performance will be done using standard tests that are routinely carried out as part of the athletes' training program in every branch of sports. For triathletes running times for 3000 meters are measured, for swimmers their times for set distances (50 meters,100 meters, 400 meters, etc). All these measures will be done without deviation from the regular training routine. Also general parameters will be measured like standing heart rate and reclining heart rate, and heart rate at awakening in the morning.

Stage 2:

At this stage the participants will be divided randomly into two groups. In the course of an additional training cycle of two weeks one group labeled 'A' will be given additional sleep time of one to two hours. The second group (group 'B') shall continue with no change. In the course of the two weeks sleep parameters of both groups will be assessed and analyzed, and athletic performance during routine training will continue to be measured and tabulated. After these two weeks the two groups will be crossed over, group 'A' will return to a routine sleep schedule, i.e. the extra sleep time will be removed and group 'B' will get additional sleep time. All the aforementioned measures will be collected during two weeks (sleep quality, athletic performance during training).

After analysis of the results further testing will be recommended as needed as well as changes in training programs, daily scheduling and sleep schedules.

During the entire study there will be close monitoring of injuries among participants. Events will be defined as injuries (according to the number of treatments by a physiotherapist or visits to a doctor) or near injuries and will be quantified, and correlations will be sought between performance, injuries and sleep duration.

In both stages in addition to wearing a heart rate belt, the participants will be asked to fill out a questionnaire before and after sleep during the entire study (see attached document).

Note: Suunto is a Finnish company that makes advanced sports watches and sensitive heart rate belts used by athletes in their training. The belt is soft, of very high quality, lightweight and contains a sensor and memory unit to store the heart rate data of the participant. It is approved for routine use for monitoring heart rate in people engaged in physical activity.

Expected benefits:

* Better understanding of the physiology associated with sleep among adolescents involved in regular, competitive physical activity.
* Improved performance by building a sleep program, optimal wakefulness and training.

ELIGIBILITY:
Inclusion Criteria:

* Age: 13-20 years old, male and female
* Generally good health
* Willingness to participate in the study
* Healthy heart rate

Exclusion Criteria:

* Arrhythmia
* Chronic or acute illness
* Unwillingness of the subject or his/her parents to participate in the study

Ages: 13 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 19 (Actual)
Dates: Start 2011-06; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Improved athletic performance: reduced swimming and running times over predefined distances with sleep extension | 12 months
  Measure the changes in performance (running and swimmimng time) as follows: for runners- time required for 3000 m distance. for swimmers- time required for 50 m, 100 m, and 400 m, at predefined heart rates.

CONTACTS AND LOCATIONS:
Overall Officials: Eyal Shargal, PhD, Principal Investigator — Wingate Institute
Locations (1):
- Wingate Institute, Netanya, Israel

REFERENCES:
- See also: Related Info — http://www.wingate.org.il